CLINICAL TRIAL: NCT02019121
Title: Dexmedetomidine and Renal Transplants
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 521455
Record Dates: First submitted 2013-11-05; First posted 2013-12-24 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigators aim to retrospectively research patients undergoing renal transplants that received dexmedetomidine perioperatively to see if dexmedetomidine use protects renal function. Investigators hope to elucidate any association between renal transplant patients and perioperative dexmedetomidine administration, these include (but are not limited to) UOP, Cr/GFR, morbidity, mortality, in hospital complications and failure rate. Investigators will research both living and cadaveric renal transplants.

ELIGIBILITY:
Inclusion Criteria: Patients greater than or equal to 18 years old that underwent renal transplant at UC Davis Medical Center -

Exclusion Criteria: Patients that did not undergo renal transplants and patients less than 18 years old will be excluded from the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 797 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Cr/GFR improvement, postoperative mortality/morbidity (within 30 days) and overall complications | 5 years

SECONDARY OUTCOMES:
Graft failure, length of hospital stay (LOS), length of ICU stay, re-admission rate, infections, pulmonary complications. | 5 years

OTHER OUTCOMES:
length of intubation time, and length of ventilation time | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Health System, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-past-experimental-treatment-with-dexmedetomidine-in-patients-with-renal-transplants-514393/